CLINICAL TRIAL: NCT04058431
Title: Examining Osteopathic Manipulation on Making a Neuropsychological Brain of Difference in Adults With Pain: A BOD Study Protocol and Rationale for a New Approach
Brief Title: Osteopathic Manipulation Makes a Neuropsychological Difference
Acronym: BOD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Responsible Party: Principal Investigator, Mireille Rizkalla, Associate Professor, Midwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MWU2761
Record Dates: First submitted 2017-04-06; First posted 2019-08-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Change; Musculoskeletal Pain
Keywords: cognitive decline; pain; osteopathic manipulative treatment
MeSH Terms: conditions — Musculoskeletal Pain; Cognitive Dysfunction; Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Osteopathic group (Experimental): Treatment will be compromised of 8 weeks of standard care plus OMT. Each physician will maintain the same patient at recurring sessions. Osteopathic treatment is performed for 30 minutes and the techniques applied are highly individualized to the patient needs (i.e., techniques are selected based on structure/function, and techniques change over time based on treatment response). In an effort to standardize treatment, we will limit the study protocol to the following designated techniques: facilitated positional release treatment, high velocity low amplitude treatment, articulatory treatment, strain-counterstrain, muscle energy treatment, myofascial release treatment, soft tissue treatment.
  Interventions: Other: Osteopathic Manipulative Treatment; Other: Control- No Intervention

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — Osteopathic manipulative treatment (OMT) is defined as the therapeutic application of manually guided forces by an osteopathic physician to improve physiologic function and/or support homeostasis that has been altered by somatic dysfunction. Somatic (body framework) dysfunction or altered function of related components is observed in the skeletal, arthrodial and myofascial structures, and their related vascular, lymphatic, and neural elements. Techniques can use a direct method where the restrictive barrier is engaged and a final activating force is applied to correct the somatic dysfunction, or an indirect method where the restrictive barrier is disengaged and the dysfunctional body part is moved away from the restrictive barrier until tissue tension is equal in one or all planes and directions
Other: Control- No Intervention — This group will refrain from getting OMT while in the study.

SUMMARY:
Patients with pain commonly experience cognitive impairment. While symptoms of pain are effectively treated with osteopathic manipulative treatment (OMT), the cognitive piece is vastly ignored. Pain-induced cognitive dysfunction can be severe and is particularly apparent in working memory and attention. There is good reason to also expect cognitive responsiveness to OMT. Previous research has already reported related psychiatric outcomes, including relief from stress, self-perception and anxiety, suggesting that OMT may produce more global effects on cortical processing than currently thought.

DETAILED DESCRIPTION:
Patients with pain commonly experience cognitive impairment. While symptoms of pain are effectively treated with osteopathic manipulative treatment (OMT), the cognitive piece is vastly ignored. Previous research has already reported related psychiatric outcomes, including relief from stress, self-perception and anxiety, suggesting that OMT may produce more global effects on cortical processing than currently thought. The current study is designed to extend previous research in several ways:

1. To describe the neuropsychological (NP) characteristics of adults with pain within an osteopathic and allopathic setting
2. To correlate NP with clinical outcomes (pain severity, number/location of osteopathic lesions)
3. To determine if OMT is associated with improved NP function.
4. To use saliva to measure cytokine concentration of IL-1β,IL-6, IL-8, TNF-α
5. To correlate cytokine concentrations with clinical outcomes (pain severity, number/location of osteopathic lesions, NP)

ELIGIBILITY:
Inclusion Criteria:

1. 40 years of age or older;
2. seeking treatment for acute or chronic pain (neck, thoracic, shoulder, back)
3. gives a positive response to the item, "Have you had thinking problems because of your pain?";
4. agree to forego extra-trial manipulation (e.g., massage, chiropractic, physical therapy);
5. Score > 23 on the Telephone Interview for Cognitive Status;
6. written informed consent.

Exclusion Criteria:

1. recent (< 2 month) or planned surgery within the duration of the study;
2. use of medication that could interfere with cytokine measurements;
3. recent (< 2 month) changes to psychotropic medication within the duration of the study;
4. history of manipulation within the past six months.
5. diagnosed neurocognitive disorders;
6. contraindication to receiving OMT.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
neuropsychology change | baseline, week 8, week 12
  standardized assessment battery
pain scale change | baseline, week 8, week 12
  1-10
inflammatory markers change | baseline, week 8, week 12
  cortisol
inflammatory marker | baseline, week 8, week 12
  TNF Alpha
Inflammatory marker | baseline, week 8, week 12
  IL 6

CONTACTS AND LOCATIONS:
Overall Officials: mireille rizkalla, phd, Principal Investigator — Midwestern University; Katrina Ivkovic, Study Director — Midwestern University
Locations (1):
- Midwestern Multispecialty Clinic, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No